CLINICAL TRIAL: NCT04860752
Title: SAPIEN 3 Ultra EU Post-Market Observational Study
Brief Title: SAPIEN 3 Ultra EU PMS
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-02
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Aortic Stenosis; Aortic Valve Stenosis
Keywords: Transcatheter aortic valve implantation (TAVI); SAPIEN 3 Ultra THV; Edwards Lifesciences
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: Yes

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Subjects will undergo TAVI

SUMMARY:
This study will evaluate real-world outcomes for the SAPIEN 3 Ultra Transcatheter Heart Valve System in transcatheter aortic valve implantation centres that are implementing minimalist periprocedural practices and facilitating early discharge home.

DETAILED DESCRIPTION:
This is a prospective, observational, single-arm, multicentre, post-market study.

ELIGIBILITY:
Inclusion Criteria:

1. Will undergo TAVI with the Edwards SAPIEN 3 Ultra System
2. Less than 80 years of age at time of the procedure
3. Low surgical risk
4. Meets clinical and procedural requirements for early discharge
5. The subject or subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent

Exclusion Criteria:

1. Medical, social, or psychological conditions that preclude appropriate consent and follow-up, including subjects under guardianship
2. Considered to be part of a vulnerable population
3. Active SARS-CoV-2 infection (Coronavirus-19 [COVID-19]) or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
4. Cannot tolerate an anticoagulation/antiplatelet regimen
5. Active bacterial endocarditis
6. Participating in a drug or device study that has not reached its primary endpoint

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who will undergo TAVI with the Edwards SAPIEN 3 Ultra System as part of standard-of-care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- Austria (3):
  - LKH-Univ. Graz Klinik, Auenbruggerplaz 15, Graz
  - Universitaetsklinikum St. Poelten, Klinik fuer Innere Medizin 3, Sankt Pölten
  - Medizinische Universitaet Vienna, Vienna
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Teiskontie 35, Tampere
- France (4):
  - Clinique St Augustin, Bordeaux
  - Institut Hospitalier Jacques Cartier Massy, Massy
  - CHU Bordeaux Hôpital Haut-Lévêque, Pessac
  - CHU Hopital Charles Nicolle Rouen, Rouen
- Germany (7):
  - Hdz Bad Oeynhausen, Bad Oeynhausen
  - Deutches Herzzentrum Berlin, Berlin
  - Universitäres Herz- und Gefäßzentrum UKE Hamburg, Hamburg
  - UKSH University Hospital Kiel, Kiel
  - Hospital Universitaet Mainz, Mainz
  - Deutsches Herzzentrum Muenchen, München
  - LMU, Klinikum der Universitaet Meunchen - Großhadern, München
- Italy (8):
  - Ospedale Moscati, Contrada Amoretta, Avellino
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Irccs Ismett, Palermo
  - Ospedale San Camillo, Roma
  - Ospedale Santissima Annunziata, Sassari
  - Ospedale Mauriziano, Torino
  - Azienda ULSS2 Marca Trevigiana, Treviso
  - Ospedale Civile Maggiore, Verona
- Oslo Universitetssykehus Rikshospitalet, Oslo, Norway
- Portugal (3):
  - Hospital de Santa Cruz, Centro Hospitalar de Lisboa Ocidental , Estrada do Forte do Alto do Duque, Lisbon
  - Hospital Santa Maria, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Spain (5):
  - Complexo Hospitalario Universitario Coruna, A Coruña
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Valdecilla Santander, Av. de Valdecilla 25, Santander
  - Hospital Alvara Cunqueiro, Estrada de Clara Campoamor 341, Vigo
- Universitatsspital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Leeds General Infirmary, Leeds
  - St Thomas' Hospital, London
  - Oxford John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcatheter Aortic Valve Implantation (TAVI): Patients receive Transcatheter Aortic Valve Implantation (TAVI)
Period: Overall Study
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Started | 500
Completed | 482
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (4.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217
  Male | 283
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Length of Index Hospitalization
Description: Number of days in hospital after the procedure
Time Frame: Discharge from hospital, expected to be within 1-5 days post-procedure
Population: As treated - all patients enrolled in the trial
Measure: Mean (Standard Error); unit: days
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 500
days | 3.3 (0.11)

2. Secondary Outcome: Death
Description: Number of patients who died
Time Frame: 1 year
Population: As treated - all patients enrolled in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 500
Participants | 9

3. Secondary Outcome: Stroke
Description: Number of patients who had a stroke
Time Frame: 1 year
Population: As treated - all patients enrolled in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 500
Participants | 7

4. Secondary Outcome: New Requirement for Permanent Pacemaker
Description: Number of patients who received a new permanent pacemaker
Time Frame: 1 year
Population: As treated - all patients enrolled in the trial who did not previously have a permanent pacemaker implanted
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 474
Participants | 51

5. Secondary Outcome: Aortic Valve Reintervention
Description: Number of patients who required valve reintervention
Time Frame: 1 year
Population: As treated - all patients enrolled in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 500
Participants | 3

6. Secondary Outcome: Aortic Regurgitation
Description: Number of patients who had moderate or greater aortic regurgitation
Time Frame: At discharge from hospital, expected to be within 1-5 days post-procedure
Population: Patients implanted with study valve who received an echocardiogram at discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 399
Participants | 2

7. Secondary Outcome: Mean Gradient
Description: Mean gradient (mmHg)
Time Frame: At discharge from hospital, expected to be within 1-5 days post-procedure
Population: Patients implanted with study valve who received an echocardiogram at discharge
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 413
mmHg | 12.8 (0.24)

8. Secondary Outcome: Effective Orifice Area
Description: Aortic valve area (cm2)
Time Frame: At discharge from hospital, expected to be within 1-5 days post-procedure
Population: Patients implanted with study valve who received an echocardiogram at discharge
Measure: Mean (Standard Error); unit: cm2
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 273
cm2 | 1.6 (0.02)

9. Secondary Outcome: Discharge Location
Description: Number of patients who were discharged to home or self-care (routine discharge)
Time Frame: At discharge from hospital, expected to be within 1-5 days post-procedure
Population: As treated - all patients enrolled in the trial
Measure: Number; unit: participants
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
Number analyzed (Participants) | 500
participants | 436

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Transcatheter Aortic Valve Implantation (TAVI)
All-Cause Mortality (participants affected / at risk) | 9/500
Serious Adverse Events (participants affected / at risk) | 157/500
Other Adverse Events (participants affected / at risk) | 42/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Aortic Valve Implantation (TAVI) (N=500)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 12 (13)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 27 (27)
Atrioventricular block first degree (Cardiac disorders) | 8 (8)
Atrioventricular block second degree (Cardiac disorders) | 11 (11)
Bradycardia (Cardiac disorders) | 2 (3)
Bundle branch block bilateral (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 15 (15)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 9 (15)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 4 (4)
Sinus node dysfunction (Cardiac disorders) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Device embolisation (General disorders) | 2 (2)
Prosthetic cardiac valve regurgitation (General disorders) | 4 (4)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cholangitis infective (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Aortic annulus rupture (Injury, poisoning and procedural complications) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 5 (5)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 7 (8)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Transvalvular pressure gradient increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 5 (5)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 5 (5)
Device deployment issue (Product Issues) | 1 (1)
Patient-device incompatibility (Product Issues) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Haematuria (Renal and urinary disorders) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal cavity drainage (Surgical and medical procedures) | 1 (2)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Hip surgery (Surgical and medical procedures) | 1 (1)
Pancreaticoduodenectomy (Surgical and medical procedures) | 1 (1)
Aortic disorder (Vascular disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (8)
Hypertension (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (5)
Peripheral artery occlusion (Vascular disorders) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Aortic Valve Implantation (TAVI) (N=500)
Bundle branch block left (Cardiac disorders) | 42 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT04860752/Prot_SAP_000.pdf